CLINICAL TRIAL: NCT03970213
Title: Effects of Intravenous Tranexamic Acid During Rhytidectomy - a Randomized, Controlled, Double-blind Pilot Study
Brief Title: Intravenous Tranexamic Acid During Rhytidectomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Glasgold Group Plastic Surgery (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: GGPS19-01
Record Dates: First submitted 2019-05-29; First posted 2019-05-31 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Bleeding; Bruising Face; Swelling Lips & Face
Keywords: Tranexamic acid; Rhytidectomy; Facelift
MeSH Terms: conditions — Hemorrhage; Facies | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Only the CRNA who is administering the medications is unmasked until completion of the data collection period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Placebo Comparator): Intravenous normal saline (50cc) given over 15 minutes starting just prior to skin incision, and repeated 4 hours later
  Interventions: Drug: Normal Saline 0.9% Infusion Solution Bag
- TXA Group (Experimental): One gram of intravenous tranexamic acid (TXA) in normal saline (50cc) given over 15 minutes starting just prior to skin incision, and repeated 4 hours later
  Interventions: Drug: Tranexamic Acid 100Mg/Ml Inj Vil 10Ml

INTERVENTIONS:
Drug: Tranexamic Acid 100Mg/Ml Inj Vil 10Ml — IV TXA given during surgery
  Arms: TXA Group
Drug: Normal Saline 0.9% Infusion Solution Bag — IV saline given during surgery
  Arms: Control Group

SUMMARY:
This is a prospective, randomized, double-blind study investigating whether intravenous tranexamic acid has any effect on rhytidectomy surgery, or the subsequent postoperative sequelae. Intraoperative bleeding and postoperative ecchymosis and edema are subjectively rated and complications are noted.

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blind pilot study investigating whether intravenous tranexamic acid has any effect on rhytidectomy surgery, or the subsequent postoperative sequelae. Intraoperative bleeding is rated on a scale of mild, moderate, or severe and given a score of 1-3. Postoperative ecchymosis and edema are subjectively rated by both patient and surgeon on postoperative days 1, 6, and 9 using a similar mild/moderate/severe scale and scored 1-3, respectively. Any surgical or postoperative complications are noted. Scores are aggregated for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing rhytidectomy surgery at Glasgold Group Plastic Surgery

Exclusion Criteria:

* History of bleeding disorder, history of thromboembolic events, history of seizure, active use of oral contraceptive pills or hormone replacement therapy, participant preference

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-05-30 (Estimated); Primary Completion 2019-08-30 (Estimated); Study Completion 2019-08-30 (Estimated)

PRIMARY OUTCOMES:
Intraoperative bleeding | Surgical time
  Subjective measure of intraoperative blood loss (mild, moderate, or severe)
Postoperative ecchymosis | Postoperative day 1
  Subjective measure of bruising rated as mild, moderate, or severe
Postoperative ecchymosis | Postoperative day 6
  Subjective measure of bruising rated as mild, moderate, or severe
Postoperative ecchymosis | Postoperative day 9
  Subjective measure of bruising rated as mild, moderate, or severe
Postoperative edema | Postoperative day 1
  Subjective measure of swelling rated as mild, moderate, or severe
Postoperative edema | Postoperative day 6
  Subjective measure of swelling rated as mild, moderate, or severe
Postoperative edema | Postoperative day 9
  Subjective measure of swelling rated as mild, moderate, or severe

SECONDARY OUTCOMES:
Postoperative hematoma/seroma | 10 days postoperative
  Documentation of any postoperative collections seen during the first 10 days following surgery
Complications | 10 days postoperative
  Documentation of any surgical or postoperative complications

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Glasgold, MD, Study Director — Glasgold Group Plastic Surgery
Locations (1):
- Glasgold Group Plastic Surgery, Princeton, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient demographics, surgical procedure performed, primary and secondary outcomes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Will be made available via publication